CLINICAL TRIAL: NCT03170544
Title: A Single Ascending Dose Clinical Trial to Study the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MK-1092 in Healthy Subjects, Subjects With Type 1 Diabetes Mellitus, and Subjects With Type 2 Diabetes Mellitus.
Brief Title: Single Ascending Dose Study of MK-1092 in Healthy Participants and in Participants With Type 1 and Type 2 Diabetes Mellitus (MK-1092-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1092-001; MK-1092-001 (Other: Merck protocol number)
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Results first posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Insulin Lispro; Glucose; Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Part 1, MK-1092, 4.0 nmol/kg (Experimental): MK-1092, 4.0 nmol/kg, SC, as a single dose under the euglycemic clamp, in healthy participants
  Interventions: Drug: MK-1092, 4.0 nmol/kg; Drug: Placebo to glargine; Other: Dextrose
- Part 1, MK-1092, 8.0 nmol/kg (Experimental): MK-1092, 8.0 nmol/kg, SC, as a single dose under the euglycemic clamp, in healthy participants
  Interventions: Drug: MK-1092, 8.0 nmol/kg; Drug: Placebo to glargine; Other: Dextrose
- Part 1, MK-1092, 16 nmol/kg (Experimental): MK-1092, 16 nmol/kg, SC, as a single dose under the euglycemic clamp, in healthy participants
  Interventions: Drug: MK-1092, 16 nmol/kg; Drug: Placebo to glargine; Other: Dextrose
- Part 1, MK-1092, 32 nmol/kg (Experimental): MK-1092, 32 nmol/kg, SC, as a single dose under the euglycemic clamp, in healthy participants
  Interventions: Drug: MK-1092, 32 nmol/kg; Drug: Placebo to glargine; Other: Dextrose
- Part 1, MK-1092, 64 nmol/kg (Experimental): MK-1092, 64 nmol/kg, SC, as a single dose under the euglycemic clamp, in healthy participants
  Interventions: Drug: MK-1092, 64 nmol/kg; Drug: Placebo to glargine; Other: Dextrose
- Part 1, Glargine, 3.0 nmol/kg (Active Comparator): Glargine, 3.0 nmol/kg, SC, as a single dose under the euglycemic clamp, in healthy participants
  Interventions: Drug: Glargine 3.0 nmol/kg; Drug: Placebo to MK-1092; Other: Dextrose
- Part 2, MK-1092, 8.0 nmol/kg + lispro, 1.2 nmol/kg (Experimental): MK-1092, 8.0 nmol/kg dose selection based on Part 1 + lispro (Humalog®), 1.2 nmol/kg, as a single dose, in healthy participants
  Interventions: Drug: MK-1092, 8.0 nmol/kg; Drug: Lispro 1.2 nmol/kg; Other: Dextrose
- Part 3, MK-1092, 8.0 nmol/kg (Experimental): MK-1092, (8.0 nmol/kg based on Part 1), SC, in participants with T1DM.
  Interventions: Drug: MK-1092, 8.0 nmol/kg; Drug: Placebo to glargine; Other: Dextrose; Biological: Insulin
- Part 3, MK-1092, 32 nmol/kg (Experimental): MK-1092, 32 nmol/kg, SC, as a single dose, in participants with T1DM
  Interventions: Drug: MK-1092, 32 nmol/kg; Drug: Placebo to glargine; Other: Dextrose; Biological: Insulin
- Part 3, Glargine, 3.0 nmol/kg (Active Comparator): Glargine, 3.0 nmol/kg, SC, as a single dose, in participants with T1DM
  Interventions: Drug: Glargine 3.0 nmol/kg; Drug: Placebo to MK-1092; Other: Dextrose; Biological: Insulin
- Part 4, MK-1092, 32 nmol/kg (Experimental): MK-1092, 32 nmol/kg, SC, as a single dose, in participants with T2DM
  Interventions: Drug: MK-1092, 32 nmol/kg; Drug: Placebo to glargine; Other: Dextrose; Biological: Insulin
- Part 4, MK-1092, 16 nmol/kg (Experimental): MK-1092, 16 nmol/kg, SC, as a single dose, in participants with T2DM
  Interventions: Drug: MK-1092, 16 nmol/kg; Drug: Placebo to glargine; Other: Dextrose; Biological: Insulin
- Part 4, MK-1092, 64 nmol/kg (Experimental): MK-1092, 64 nmol/kg, SC, as a single dose, in participants with T2DM
  Interventions: Drug: MK-1092, 64 nmol/kg; Drug: Placebo to glargine; Other: Dextrose; Biological: Insulin
- Part 4, Glargine, 3.0 nmol/kg (Active Comparator): Glargine, 3.0 nmol/kg, SC, as a single dose, in participants with T2DM
  Interventions: Drug: Glargine 3.0 nmol/kg; Drug: Placebo to MK-1092; Other: Dextrose; Biological: Insulin

INTERVENTIONS:
Drug: MK-1092, 4.0 nmol/kg — MK-1092, 4.0 nmol/kg, SC, as a single dose under the euglycemic clamp, in participants
  Arms: Part 1, MK-1092, 4.0 nmol/kg
Drug: MK-1092, 8.0 nmol/kg — MK-1092, 8.0 nmol/kg, SC, as a single dose under the euglycemic clamp, in participants
  Arms: Part 1, MK-1092, 8.0 nmol/kg; Part 2, MK-1092, 8.0 nmol/kg + lispro, 1.2 nmol/kg; Part 3, MK-1092, 8.0 nmol/kg
Drug: MK-1092, 16 nmol/kg — MK-1092, 16 nmol/kg, SC, as a single dose under the euglycemic clamp, in participants
  Arms: Part 1, MK-1092, 16 nmol/kg; Part 4, MK-1092, 16 nmol/kg
Drug: MK-1092, 32 nmol/kg — MK-1092, 32 nmol/kg, SC, as a single dose under the euglycemic clamp, in participants
  Arms: Part 1, MK-1092, 32 nmol/kg; Part 3, MK-1092, 32 nmol/kg; Part 4, MK-1092, 32 nmol/kg
Drug: MK-1092, 64 nmol/kg — MK-1092, 64 nmol/kg, SC, as a single dose under the euglycemic clamp, in participants
  Arms: Part 1, MK-1092, 64 nmol/kg; Part 4, MK-1092, 64 nmol/kg
Drug: Glargine 3.0 nmol/kg — Glargine 3.0 nmol/kg, SC, as a single dose
  Arms: Part 1, Glargine, 3.0 nmol/kg; Part 3, Glargine, 3.0 nmol/kg; Part 4, Glargine, 3.0 nmol/kg
Drug: Lispro 1.2 nmol/kg — Lispro (Humalog®), 1.2 nmol/kg, IV infusion SC over 3 hours as a single dose starting ~12 hours after MK-1092 administration.
  Other Names: Humalog®
  Arms: Part 2, MK-1092, 8.0 nmol/kg + lispro, 1.2 nmol/kg
Drug: Placebo to glargine — Placebo to glargine, SC, as a single dose
  Arms: Part 1, MK-1092, 16 nmol/kg; Part 1, MK-1092, 32 nmol/kg; Part 1, MK-1092, 4.0 nmol/kg; Part 1, MK-1092, 64 nmol/kg; Part 1, MK-1092, 8.0 nmol/kg; Part 3, MK-1092, 32 nmol/kg; Part 3, MK-1092, 8.0 nmol/kg; Part 4, MK-1092, 16 nmol/kg; Part 4, MK-1092, 32 nmol/kg; Part 4, MK-1092, 64 nmol/kg
Drug: Placebo to MK-1092 — Placebo to MK-1092, SC, as a single dose
  Arms: Part 1, Glargine, 3.0 nmol/kg; Part 3, Glargine, 3.0 nmol/kg; Part 4, Glargine, 3.0 nmol/kg
Other: Dextrose — 20% solution for continuous infusion for the duration of the glucose clamp as needed to maintain blood sugar at pre-clamp target levels.
  Other Names: Glucose
Biological: Insulin — Participants will receive insulin IV, as needed, prior to dosing and clamp initiation and after dosing.
  Arms: Part 3, Glargine, 3.0 nmol/kg; Part 3, MK-1092, 32 nmol/kg; Part 3, MK-1092, 8.0 nmol/kg; Part 4, Glargine, 3.0 nmol/kg; Part 4, MK-1092, 16 nmol/kg; Part 4, MK-1092, 32 nmol/kg; Part 4, MK-1092, 64 nmol/kg

SUMMARY:
This is an active- and placebo-controlled, single-site, four-part trial of MK-1092 in healthy adult participants, in participants with type 1 diabetes mellitus (T1DM), and in participants with type 2 diabetes mellitus (T2DM). The primary hypothesis for this study is that at a dose with sufficient safety, the mean maximal glucose infusion rate (GIRmax) after single subcutaneous (SC) administration of MK-1092 in adult participants with T1DM is within an acceptable range. (Part 3)

DETAILED DESCRIPTION:
There will be 4 parts in this study. In Part 1, healthy adult participants will be randomized to receive blinded MK-1092 subcutaneously (SC) or glargine SC, as a single dose under the euglycemic clamp. Once a safe and tolerated dose that achieves GIRmax is identified in Part 1, Part 2 will start. In Part 2, 4 different healthy adult participants will be enrolled in a single panel and receive open-label MK-1092 SC as a single dose under the euglycemic clamp and also receive an intravenous infusion of Humalog®. In Part 3, adult participants with T1DM will be randomized to receive blinded MK-1092 SC or insulin glargine SC, as a single dose under the euglycemic clamp. Part 4 includes a 3-period (Periods 1, 2, and 3) design that will explore up to 3 single subcutaneous doses of MK-1092 or insulin glargine in participants with Type 2 diabetes mellitus.

ELIGIBILITY:
Subject Inclusion Criteria

All participants

* Be a healthy male, or healthy female participant (excluding diabetes mellitus in Part 3 participants) of non-child bearing potential. A female non-child bearing potential is one who is postmenopausal without menses for at least 1 year or whose status is post hysterectomy, bilateral oophorectomy, or tubal ligation.
* Be judged to be in good health based on medical history, physical exam, vital sign measurements, electrocardiogram (ECG) and laboratory safety tests
* Have adequate venous access to support execution of trial procedures

For Parts 1 and 2 (Healthy adult participants)

* Healthy male and female participants between the ages of 18 and 50 years (inclusive)
* Have a Body Mass Index (BMI) ≥18.5 kg/m^2 and ≤28.0 kg/m^2 at screening
* Have fasting blood glucose values at screening must be <100 mg/dL
* Be a non-smoker and/or has not used nicotine or nicotine-containing products (e.g., nicotine patch) for at least approximately 3 months.

For Part 3 (Adult participants with T1DM):

* Be male, or female of non-childbearing potential between 18 to 60 years of age
* Have a diagnosis of T1DM as defined by standard diagnostic criteria for ≥12 months at time of the pretrial (screening) visit
* Have a BMI ≥18.5 kg/m^2 and ≤32 kg/m^2 at screening.
* Be on stable doses of basal insulin over the 2-week period prior to screening and over the 2 weeks prior to dosing
* Have a total daily insulin requirement (basal plus prandial) of ≤1.2 units/kg at screening
* Have a hemoglobin A1C (HbA1c) ≤10% at the screening visit.
* Be a non-smoker or smoker who uses no more than 5 cigarettes or equivalent (e.g., e-cigarettes) per day over the prior 3-month period also may be enrolled (at the discretion of the investigator).
* Have a serum C-peptide concentration ≤0.7 ng/mL with a concurrent plasma glucose >90 mg/dL at screening or anytime within 24 weeks prior to screening.

For Part 4 (Adult participants with T2DM):

* Diagnosis of T2DM as defined by standard diagnostic criteria for ≥12 months at time of pretrial screening.
* Have a BMI ≥18.5 kg/m2 and ≤35.0 kg/m^2 at screening. BMI = mass (kg)/height (m)^2.
* Have a hemoglobin A1C (HbA1c) ≥6.5% and ≤10.0%.
* T2DM participants are not required to have been on insulin. If using insulin as background therapy, subjects should have a total daily insulin requirement of ≤1.2 units/kg, and have been on stable doses of basal insulin over the 2-week period prior to screening and over the 2 weeks prior to dosing.
* Be a non-smoker or smoker who uses no greater than 5 cigarettes or equivalent (e.g., e-cigarettes) daily over the prior 3-month period.

Subject Exclusion Criteria

All participants

* Is mentally or legally incapacitated
* Has a history of clinically significant endocrine (excluding diabetes mellitus in Part 3 participants), gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary or major neurological (including stroke and chronic seizures) abnormalities or diseases.
* Has a systolic blood pressure (SBP) ≥140 mm Hg and/or a diastolic blood pressure (DBP) ≥90 mm Hg at screening.
* Is positive for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV) at screening.
* Has a history of cancer (malignancy) Exceptions: (1) Participants with adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix may participate in the trial; (2) Participants with other malignancies which have been successfully treated ≥10 years prior to the pretrial (screening) visit
* Has a history of significant multiple and/or severe allergies (e.g. food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability (i.e. systemic allergic reaction) to prescription or non-prescription drugs or food.
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the pretrial (screening) visit.
* Has participated in another investigational trial within 4 weeks.
* Has been randomized to, and received MK-5160 in prior clinical studies.
* Has a QTcF interval >450 msec, has a history of risk factors for Torsades de Pointes (e.g., heart failure/cardiomyopathy or family history of Long QT Syndrome).
* Has uncorrected hypokalemia
* Has uncorrected hypomagnesemia
* Is taking concomitant medications that prolong the QT/QTc interval.
* Is unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies beginning approximately 2 weeks prior to administration of the initial dose of trial drug, throughout the trial, until the post-trial visit.
* Has had a vaccination within 12 weeks of the pretrial visit.
* Consumes greater than 3 glasses of alcoholic beverages per day.
* Consumes excessive amounts, defined as greater than 6 servings caffeinated beverages per day.
* Is currently a regular or recreational user of cannabis, any illicit drugs or has a history of drug (including alcohol) abuse within approximately 6 months
* Has used systemic (intravenous, oral, inhaled) glucocorticoids within 3 months of screening or is anticipated to require treatment with systemic glucocorticoids during study participation.

For Part 1 and Part 2 (Healthy Adult Participants)

- Has an estimated creatinine clearance of <90 mL/min based on Cockcroft-Gault equation

For Part 3 (Adult participants with T1DM):

* Has a history of diabetic ketoacidosis in the last 6 months prior to screening.
* Has an estimated creatinine clearance of <60 mL/min based on the Cockcroft-Gault equation at screening
* Has the diagnosis of hypoglycemia unawareness, or has had one or more severe hypoglycemic episodes associated with hypoglycemic seizures, comas or unconsciousness within 6 months prior to dosing.
* Has other major medical problems requiring medication (i.e., history of myocardial infarction (MI), hypercholesterolemia).
* Has a known history of celiac disease or significant food allergy, at the discretion of the investigator and Sponsor.
* Has a history of hypersensitivity to pharmacologic insulins or to any of the inactive ingredients in recombinant human insulin, or to any E.coli-derived drug product.

For Part 4 (Adult participants with T2DM):

* Participant has an estimated creatinine clearance of <60 mL/min based on the Cockcroft-Gault equation.
* Has a history of diabetic ketoacidosis in the last 6 months prior to screening.
* Has the diagnosis of hypoglycemia unawareness, or has had one or more severe hypoglycemic episodes associated with hypoglycemic seizures, comas or unconsciousness within 6 months prior to dosing.
* Has a known history of celiac disease or significant food allergy, at the discretion of the Investigator and Sponsor.
* Has been treated with a thiazolidinedione or injectable non-insulin anti-diabetic therapy within the past three months prior to dosing.
* Has a history of hypersensitivity to pharmacologic insulins or to any of the inactive ingredients in regular human insulin, or to any E.coli-derived drug product.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- ProSciento Inc. ( Site 0001), Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Walford GA, Duncan KE, Hernandez M, Vaddady P, Hompesch M, Morrow L, Stoch SA. A Randomized, Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of a Novel Insulin Dimer. Clin Pharmacol Ther. 2022 Jul;112(1):125-132. doi: 10.1002/cpt.2607. Epub 2022 May 3. PMID 35390172

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 4-part study, participants received MK-1092 or glargine: Part 1 - healthy adult participants; Part 2, healthy adult participants received MK-1092 and also insulin lispro (Humalog®); Part 3 - adult participants with Type 1 diabetes mellitus; Part 4 had 3 periods (Periods 1, 2, and 3), participants with Type 2 diabetes mellitus.
Groups:
- Part 1 (Healthy Adults) Glargine 3.0 Nmol/kg: Glargine, 3.0 nmol/kg, SC, as a single dose under the euglycemic clamp in healthy participants
- Part 1 (Healthy Adults) MK-1092 4.0 Nmol/kg: MK-1092, 4.0 nmol/kg, SC, as a single dose under the euglycemic clamp in healthy participants
- Part 1 (Healthy Adults) MK-1092 8.0 Nmol/kg: MK-1092, 8.0 nmol/kg, SC, as a single dose under the euglycemic clamp in healthy participants
- Part 1 (Healthy Adults) MK-1092 16 Nmol/kg: MK-1092, 16 nmol/kg, SC, as a single dose under the euglycemic clamp in healthy participants
- Part 1 (Healthy Adults) MK-1092 32 Nmol/kg: MK-1092, 32 nmol/kg, SC, as a single dose under the euglycemic clamp in healthy participants
- Part 1 (Healthy Adults) MK-1092 64 Nmol/kg: MK-1092, 64 nmol/kg, SC, as a single dose under the euglycemic clamp in healthy participants
- Part 2 (Healthy Adults) MK-1092 + Insulin Lipro: MK-1092 8 nmol/kg SC+ Insulin Lipro (Humalog®) 1.2 nmol/kg IV, as a single dose under the euglycemic clamp in healthy participants
- Part 3 (T1DM) Glargine 3.0 Nmol/kg: Glargine, 3.0 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with T1DM
- Part 3 (T1DM) MK-1092 8.0 Nmol/kg: MK-1092 SC 8.0 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with T1DM
- Part 3 (T1DM) MK-1092 32 Nmol/kg: MK-1092 SC 32 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with T1DM
- Part 4 (T2DM) Glargine: Glargine, SC, 3.0 nmol/kg, as a single dose in Periods 1, 2, and 3 under the euglycemic clamp in participants with T2DM
- Part 4 (T2DM) MK-1092: MK-1092, SC, 32-, 16-, and 64 nmol/kg in Periods 1, 2, and 3, respectively, as a single dose under the euglycemic clamp in participants with T2DM
Period: Part 1
Arm/Group | Part 1 (Healthy Adults) Glargine 3.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 4.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 8.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 16 Nmol/kg | Part 1 (Healthy Adults) MK-1092 32 Nmol/kg | Part 1 (Healthy Adults) MK-1092 64 Nmol/kg | Part 2 (Healthy Adults) MK-1092 + Insulin Lipro | Part 3 (T1DM) Glargine 3.0 Nmol/kg | Part 3 (T1DM) MK-1092 8.0 Nmol/kg | Part 3 (T1DM) MK-1092 32 Nmol/kg | Part 4 (T2DM) Glargine | Part 4 (T2DM) MK-1092
Started | 10 | 6 | 6 | 7 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 9 | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Not treated | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 1 (Healthy Adults) Glargine 3.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 4.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 8.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 16 Nmol/kg | Part 1 (Healthy Adults) MK-1092 32 Nmol/kg | Part 1 (Healthy Adults) MK-1092 64 Nmol/kg | Part 2 (Healthy Adults) MK-1092 + Insulin Lipro | Part 3 (T1DM) Glargine 3.0 Nmol/kg | Part 3 (T1DM) MK-1092 8.0 Nmol/kg | Part 3 (T1DM) MK-1092 32 Nmol/kg | Part 4 (T2DM) Glargine | Part 4 (T2DM) MK-1092
Started | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3
Arm/Group | Part 1 (Healthy Adults) Glargine 3.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 4.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 8.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 16 Nmol/kg | Part 1 (Healthy Adults) MK-1092 32 Nmol/kg | Part 1 (Healthy Adults) MK-1092 64 Nmol/kg | Part 2 (Healthy Adults) MK-1092 + Insulin Lipro | Part 3 (T1DM) Glargine 3.0 Nmol/kg | Part 3 (T1DM) MK-1092 8.0 Nmol/kg | Part 3 (T1DM) MK-1092 32 Nmol/kg | Part 4 (T2DM) Glargine | Part 4 (T2DM) MK-1092
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 6 | 6 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 6 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 4
Arm/Group | Part 1 (Healthy Adults) Glargine 3.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 4.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 8.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 16 Nmol/kg | Part 1 (Healthy Adults) MK-1092 32 Nmol/kg | Part 1 (Healthy Adults) MK-1092 64 Nmol/kg | Part 2 (Healthy Adults) MK-1092 + Insulin Lipro | Part 3 (T1DM) Glargine 3.0 Nmol/kg | Part 3 (T1DM) MK-1092 8.0 Nmol/kg | Part 3 (T1DM) MK-1092 32 Nmol/kg | Part 4 (T2DM) Glargine | Part 4 (T2DM) MK-1092
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis set included all randomized and treated participants.
Groups:
- Part 1 (Healthy Adults) MK-1092 16 Nmol/kg: MK-1092, 16 nmol/kg, SC, as a single dose under the euglycemic clamp, in healthy participants
- Part 2 (Healthy Adults) MK-1092 + Insulin Lipro Humalog: MK-1092 8 nmol/kg SC+ Insulin Lipro (Humalog®) 1.2 nmol/kg IV, as a single dose under the euglycemic clamp in healthy participants
- Part 3 (T1DM) MK-1092 8.0 Nmol/kg: MK-1092 8 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with T1DM
- Part 3 (T1DM) MK-1092 32 Nmol/kg: MK-1092 32 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with T1DM
- Total: Total of all reporting groups
Arm/Group | Part 1 (Healthy Adults) Glargine 3.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 4.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 8.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 16 Nmol/kg | Part 1 (Healthy Adults) MK-1092 32 Nmol/kg | Part 1 (Healthy Adults) MK-1092 64 Nmol/kg | Part 2 (Healthy Adults) MK-1092 + Insulin Lipro Humalog | Part 3 (T1DM) Glargine 3.0 Nmol/kg | Part 3 (T1DM) MK-1092 8.0 Nmol/kg | Part 3 (T1DM) MK-1092 32 Nmol/kg | Part 4 (T2DM) Glargine | Part 4 (T2DM) MK-1092 | Total
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 4 | 4 | 6 | 6 | 3 | 6 | 69
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.3 (8.5) | 37.5 (12.0) | 33.5 (9.1) | 34.2 (8.7) | 35.2 (9.3) | 35.0 (5.7) | 45.3 (2.6) | 39.0 (12.0) | 34.2 (10.0) | 40.0 (10.4) | 52.0 (9.6) | 51.5 (4.3) | 38.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 3 | 9
  Male | 10 | 5 | 6 | 6 | 6 | 6 | 2 | 4 | 6 | 4 | 2 | 3 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 2 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 5 | 19
  Not Hispanic or Latino | 9 | 3 | 4 | 3 | 6 | 5 | 3 | 4 | 6 | 6 | 0 | 1 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 1 | 0 | 1 | 3 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 15
  White | 4 | 5 | 6 | 4 | 3 | 5 | 2 | 4 | 5 | 4 | 3 | 6 | 51
  More than one race | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An adverse event is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. Adverse events that occurred beyond 14 days of dosing were considered Post-Trial AEs. Given the half-life of MK-1092 and glargine, any events observed beyond 14 days would not be considered a result of study drug and were therefore presented together.
Time Frame: Up to 112 days
Population: The analysis population included all participants who received at least one dose of the investigational drug. Post-trial adverse events were pooled across treatment groups in each part of the study.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 (Healthy Adults) Post-trial: Glargine or MK-1092 as a single dose under the euglycemic clamp in healthy participants in the Post-trial period
- Part 2 (Healthy Adults) MK-1092 + Insulin Lipro: MK-1092, 8.0 nmol/kg dose selection based on Part 1 + Insulin lipro (Humalog®), 1.2 nmol/kg, as a single dose under the euglycemic clamp in healthy participants
- Part 2 (Healthy Adults) MK-1092 + Insulin Lipro Post-Trial: MK-1092, 8.0 nmol/kg dose selection based on Part 1 + Insulin lipro (Humalog®), 1.2 nmol/kg, as a single dose under the euglycemic clamp in healthy participants in the Post-trial period
- Part 3 (T1DM) MK-1092 8.0 Nmol/kg: MK-1092, (8.0 nmol/kg based on Part 1), SC, as a single dose under the euglycemic clamp in participants with T1DM.
- Part 3 (T1DM) MK-1092 32 Nmol/kg: MK-1092, 32 nmol/kg, SC, as a single dose, in participants with T1DM
- Part 3 (T1DM) Post-Trial: Glargine or MK-1092 as a single dose under the euglycemic clamp in participants with T1DM in the Post-trial period
- Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 1): Glargine, 3.0 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with T2DM in Period 1
- Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 2): Glargine, 3.0 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with T2DM in Period 2
- Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 3): Glargine, 3.0 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with T2DM in Period 3
- Part 4 (T2DM) MK-1092 32 Nmol/kg (Period 1): MK-1092, 32 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with T2DM
- Part 4 (T2DM) MK-1092 16 Nmol/kg (Period 2): MK-1092, 16 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with T2DM
- Part 4, (T2DM) MK-1092 64 Nmol/kg (Period 3): MK-1092, 64 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with T2DM
- Part 4 (T2DM) Post-Trial: Glargine or MK-1092 as a single dose under the euglycemic clamp in participants with T2DM in the Post-trial period
Arm/Group | Part 1 (Healthy Adults) Glargine 3.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 4.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 8.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 16 Nmol/kg | Part 1 (Healthy Adults) MK-1092 32 Nmol/kg | Part 1 (Healthy Adults) MK-1092 64 Nmol/kg | Part 1 (Healthy Adults) Post-trial | Part 2 (Healthy Adults) MK-1092 + Insulin Lipro | Part 2 (Healthy Adults) MK-1092 + Insulin Lipro Post-Trial | Part 3 (T1DM) Glargine 3.0 Nmol/kg | Part 3 (T1DM) MK-1092 8.0 Nmol/kg | Part 3 (T1DM) MK-1092 32 Nmol/kg | Part 3 (T1DM) Post-Trial | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 1) | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 2) | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 3) | Part 4 (T2DM) MK-1092 32 Nmol/kg (Period 1) | Part 4 (T2DM) MK-1092 16 Nmol/kg (Period 2) | Part 4, (T2DM) MK-1092 64 Nmol/kg (Period 3) | Part 4 (T2DM) Post-Trial
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 40 | 4 | 4 | 4 | 6 | 6 | 16 | 3 | 3 | 3 | 6 | 6 | 6 | 9
Participants | 1 | 1 | 4 | 3 | 3 | 2 | 0 | 3 | 1 | 2 | 6 | 5 | 2 | 3 | 1 | 0 | 3 | 3 | 4 | 0

2. Primary Outcome: Number of Participants Who Discontinued the Study Due to an AE
Description: as for outcome 1
Time Frame: Up to 58 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Part 3 (T1DM) Glargine 3.0 Nmol/kg: Glargine, 3.0 nmol/kg, SC, as a single dose, in participants with T1DM
- Part 3 (T1DM) MK-1092 8.0 Nmol/kg: MK-1092, (8.0 nmol/kg based on Part 1), SC, in participants with T1DM.
- Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 1): Glargine, 3.0 nmol/kg, SC, as a single dose in participants with T2DM in Period 1
- Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 2): Glargine, 3.0 nmol/kg, SC, as a single dose in participants with T2DM in Period 2
- Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 3): Glargine, 3.0 nmol/kg, SC, as a single dose, in participants with T2DM in Period 3
- Part 4 (T2DM) MK-1092 32 Nmol/kg (Period 1): MK-1092, 32 nmol/kg, SC, as a single dose, in participants with T2DM
- Part 4 (T2DM) MK-1092 16 Nmol/kg (Period 2): MK-1092, 16 nmol/kg, SC, as a single dose, in participants with T2DM
- Part 4, (T2DM) MK-1092 64 Nmol/kg (Period 3): MK-1092, 64 nmol/kg, SC, as a single dose, in participants with T2DM
Arm/Group | Part 1 (Healthy Adults) Glargine 3.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 4.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 8.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 16 Nmol/kg | Part 1 (Healthy Adults) MK-1092 32 Nmol/kg | Part 1 (Healthy Adults) MK-1092 64 Nmol/kg | Part 1 (Healthy Adults) Post-trial | Part 2 (Healthy Adults) MK-1092 + Insulin Lipro | Part 2 (Healthy Adults) MK-1092 + Insulin Lipro Post-Trial | Part 3 (T1DM) Glargine 3.0 Nmol/kg | Part 3 (T1DM) MK-1092 8.0 Nmol/kg | Part 3 (T1DM) MK-1092 32 Nmol/kg | Part 3 (T1DM) Post-Trial | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 1) | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 2) | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 3) | Part 4 (T2DM) MK-1092 32 Nmol/kg (Period 1) | Part 4 (T2DM) MK-1092 16 Nmol/kg (Period 2) | Part 4, (T2DM) MK-1092 64 Nmol/kg (Period 3) | Part 4 (T2DM) Post-Trial
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 40 | 4 | 4 | 4 | 6 | 6 | 16 | 3 | 3 | 3 | 6 | 6 | 6 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: GIRmax After a Single Dose Administration of Subcutaneous MK-1092 or Glargine to Healthy Adult Participants (Part 1)
Description: The GIRmax required to maintain blood glucose at each participants' individual clamp target, following administration of MK-1092 SC or glargine SC was determined by use of a continuous glucose infusion during the euglycemic clamp so that glucose levels remained in the euglycemic range and hypoglycemia was prevented. Blood glucose was monitored frequently (~every 5 minutes), allowing rapid changes to the rate of glucose infusion. Mean and 95% CI were based on a linear fixed effects model containing a fixed effect for treatment (MK-1092 doses, Glargine). In Part 1, 10 participants (across 5 dosing panels) received glargine. These 10 participants in Part 1 were analyzed together given the small numbers and same treatment (same dose of glargine) received.
Time Frame: Up to approximately 24 hours post-dose
Population: The analysis population included participants in Part 1 who complied with the protocol sufficiently to ensure that these data likely exhibited the effects of treatment. Compliance included exposure to treatment, availability of measurements, and absence of major protocol deviations. The glargine-treated group was pooled; n=2 participants per panel.
Measure: Mean (95% Confidence Interval); unit: mg/kg/min
Arm/Group | Part 1 (Healthy Adults) MK-1092 4.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 8.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 16 Nmol/kg | Part 1 (Healthy Adults) MK-1092 32 Nmol/kg | Part 1 (Healthy Adults) MK-1092 64 Nmol/kg | Part 1 (Healthy Adults) Glargine 3.0 Nmol/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
mg/kg/min | 0.92 [0.20 to 1.64] | 1.69 [0.97 to 2.41] | 3.10 [2.38 to 3.82] | 3.32 [2.60 to 4.04] | 4.39 [3.67 to 5.11] | 2.72 [2.16 to 3.28]

4. Primary Outcome: GIRmax After a Single Dose Administration of Subcutaneous MK-1092 or Glargine to Adult Participants With Type 1 Diabetes Mellitus (T1DM) (Part 3)
Description: The GIRmax required to maintain blood glucose at each participants' individual clamp target, following administration of MK-1092 SC or glargine SC was determined by use of a continuous glucose infusion during the euglycemic clamp so that glucose levels remained in the euglycemic range and hypoglycemia was prevented. Blood glucose was monitored frequently (~every 5 minutes), allowing rapid changes to the rate of glucose infusion. Mean and 95% CI were based on a linear fixed effects model containing a fixed effect for treatment (MK-1092 Doses, Glargine). In Part 3, 4 participants (across 2 dosing panels) received glargine. These 4 participants were analyzed together given the small numbers and the same treatment (same dose of glargine) received.
Time Frame: Up to approximately 24 hours post-dose
Population: The analysis population included participants in Part 3 who complied with the protocol sufficiently to ensure that data were likely to exhibit the effects of treatment. Compliance included exposure to treatment, availability of measurements, and absence of major protocol deviations. The glargine-treated group was pooled; n=2 participants per panel.
Measure: Mean (95% Confidence Interval); unit: mg/kg/min
Groups:
- Part 3 (T1DM) MK-1092 8.0 Nmol/kg: MK-1092, 8.0 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with Type 1 diabetes mellitus
- Part 3 (T1DM) MK-1092 32 Nmol/kg: MK-1092, 32 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with Type 1 diabetes mellitus
Arm/Group | Part 3 (T1DM) MK-1092 8.0 Nmol/kg | Part 3 (T1DM) MK-1092 32 Nmol/kg | Part 3 (T1DM) Glargine 3.0 Nmol/kg
Number analyzed (Participants) | 6 | 6 | 4
mg/kg/min | 1.33 [0.63 to 2.04] | 2.74 [2.03 to 3.44] | 2.32 [1.45 to 3.18]
Statistical Analysis 1: Comparison: Part 3 (T1DM) MK-1092 8.0 Nmol/kg; Test type: Other; Mean = 1.33, 95% CI 2-sided [0.63 to 2.04], Standard Error of Mean 0.326 — Mean (SE) and 95% CI were based on a linear fixed effects model containing a fixed effect for treatment (MK1092 Doses, Glargine); The primary hypothesis would be supported if the Bayesian posterior probability of the true mean of GIRmax of MK-1092 lying within 1.5 and 4.5 mg/kg/min exceeded the prespecified threshold of 70% (in Part 3)
Statistical Analysis 2: Comparison: Part 3 (T1DM) MK-1092 32 Nmol/kg; Test type: Other; Mean = 2.74, 95% CI 2-sided [2.03 to 3.44], Standard Error of Mean 0.326 — [estimate comment as in outcome 4, analysis 1]; [other analysis details as in outcome 4, analysis 1]

5. Secondary Outcome: GIRmax After a Single Dose Administration of Subcutaneous MK-1092 or Glargine to Adult Participants With Type 2 Diabetes Mellitus (T2DM) (Part 4)
Description: The GIRmax, following administration of MK-1092 SC or glargine SC, was determined by use of a continuous glucose infusion during the euglycemic clamp so that glucose levels remained in the euglycemic range and hypoglycemia was prevented. Blood glucose was monitored frequently (~every 5 minutes), allowing rapid changes to the rate of glucose infusion. For Part 4, a linear mixed effects model containing a fixed effect for treatment (MK-1092, Glargine), a nested effect from participants within treatment, an interaction between treatment and period (treatment by period: Period = Period 1, 2, 3) and a random effect due to participants was used. MK-1092 was administered to a single cohort of participants in Periods 1, 2, and 3. Glargine was administered to a single cohort of participants as 3.0 nmol/kg SC in Periods 1, 2, and 3.
Time Frame: Up to approximately 24 hours post-dose
Population: The analysis population included participants in Part 4 who complied with the protocol sufficiently to ensure that these data were likely to exhibit the effects of treatment, according to the underlying scientific model. Compliance included exposure to treatment, availability of measurements, and absence of major protocol deviations.
Measure: Mean (95% Confidence Interval); unit: mg/kg/min
Groups:
- Part 4 (T2DM) MK-1092 64 Nmol/kg SC (Period 3): MK-1092, 64 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with T2DM
- Part 4 (T2DM) Glargine 3.0 Nmol/kg SC (Period 1); Part 4 (T2DM) Glargine 3.0 Nmol/kg SC (Period 2): Glargine 3.0 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with T2DM
- Part 4 (T2DM) Glargine 3.0 Nmol/kg SC (Period 3): Glargine 3.0 nmol/kg, SC, as a single dose under the euglycemic clamp, in participants with T2DM
Arm/Group | Part 4 (T2DM) MK-1092 32 Nmol/kg (Period 1) | Part 4 (T2DM) MK-1092 16 Nmol/kg (Period 2) | Part 4 (T2DM) MK-1092 64 Nmol/kg SC (Period 3) | Part 4 (T2DM) Glargine 3.0 Nmol/kg SC (Period 1) | Part 4 (T2DM) Glargine 3.0 Nmol/kg SC (Period 2) | Part 4 (T2DM) Glargine 3.0 Nmol/kg SC (Period 3)
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 3 | 3
mg/kg/min | 1.90 [1.46 to 2.35] | 1.40 [0.95 to 1.84] | 2.83 [2.38 to 3.27] | 0.93 [0.30 to 1.56] | 1.43 [0.79 to 2.06] | 1.20 [0.57 to 1.83]

6. Secondary Outcome: Time-Weighted Average GIR (TWA[GIR]) After a Single Dose Administration of Subcutaneous MK-1092 or Glargine to Healthy Adult Participants (Part 1)
Description: The GIRmax required to maintain blood glucose at each participants' individual clamp target, following administration of MK-1092 SC or glargine SC was determined by use of a continuous glucose infusion during the euglycemic clamp so that glucose levels remained in the euglycemic range and hypoglycemia was prevented. Blood glucose was monitored frequently (~every 5 minutes), allowing rapid changes to the rate of glucose infusion in Part 1 only. TWA(GIR)= Time-weighted average based on GIR values calculated as AUC (area under the curve) based on GIR values observed from time zero to t divided by t, t= 24 hours. Mean and 95% CI are based on a linear fixed effects model containing a fixed effect for treatment (MK-1092 Doses, Glargine). In Part 1, 10 participants (across 5 dosing panels) received glargine. These 10 participants in Part 1 were analyzed together given the small numbers and same treatment (same dose of glargine) received.
Time Frame: Up to approximately 24 hours post-dose
Population: The analysis population included participants in Part 1 who complied with the protocol sufficiently to ensure that data were likely to exhibit the effects of treatment. Compliance included exposure to treatment, availability of measurements, and absence of major protocol deviations. The glargine-treated group was pooled; n=2 participants per panel.
Measure: Mean (95% Confidence Interval); unit: mg/kg/min
Arm/Group | Part 1 (Healthy Adults) MK-1092 4.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 8.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 16 Nmol/kg | Part 1 (Healthy Adults) MK-1092 32 Nmol/kg | Part 1 (Healthy Adults) MK-1092 64 Nmol/kg | Part 1 (Healthy Adults) Glargine 3.0 Nmol/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
mg/kg/min | 0.49 [0.00 to 0.99] | 0.97 [0.47 to 1.47] | 2.02 [1.52 to 2.52] | 1.97 [1.47 to 2.47] | 2.87 [2.37 to 3.37] | 1.70 [1.32 to 2.09]

7. Secondary Outcome: Time-Weighted Average GIR (TWA[GIR]) After a Single Dose Administration of Subcutaneous MK-1092 or Glargine to Adult Participants With T1DM (Part 3)
Description: The GIRmax required to maintain blood glucose at each participants' individual clamp target, following administration of MK-1092 SC or glargine SC was determined by use of a continuous glucose infusion during the euglycemic clamp so that glucose levels remained in the euglycemic range and hypoglycemia was prevented. Blood glucose was monitored frequently (~every 5 minutes), allowing rapid changes to the rate of glucose infusion in Part 3 only. TWA(GIR)= Time-weighted average based on GIR values calculated as AUC (area under the curve) based on GIR values observed from time zero to t divided by t, t= 24 hours. Mean and 95% CI are based on a linear fixed effects model containing a fixed effect for treatment (MK-1092 Doses, Glargine). In Part 3, 4 participants (across 2 dosing panels) received glargine. These 4 participants were analyzed together given the small numbers and same treatment (same dose of glargine) received.
Time Frame: Up to approximately 24 hours post-dose
Population: The analysis population included participants in Part 3 who complied with the protocol sufficiently to ensure that data were likely to exhibit the effects of treatment. Compliance included exposure to treatment, availability of measurements, absence of major protocol deviations. The glargine treatment group was pooled (n=2 participants per panel).
Measure: Mean (95% Confidence Interval); unit: mg/kg/min
Groups:
- Part 3 (T1DM) MK-1092 8.0 Nmol/kg: MK-1092, 8.0 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with T1DM
- Part 3 (T1DM) MK-1092 32 Nmol/kg: MK-1092, 32 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with T1DM
Arm/Group | Part 3 (T1DM) MK-1092 8.0 Nmol/kg | Part 3 (T1DM) MK-1092 32 Nmol/kg | Part 3 (T1DM) Glargine 3.0 Nmol/kg
Number analyzed (Participants) | 6 | 6 | 4
mg/kg/min | 0.72 [0.18 to 1.27] | 1.92 [1.38 to 2.46] | 1.18 [0.52 to 1.85]

8. Secondary Outcome: Time-Weighted Average GIR (TWA[GIR]) After a Single Dose Administration of Subcutaneous MK-1092 or Glargine to Adult Participants With T2DM (Part 4)
Description: The GIRmax required to maintain blood glucose at each participants' individual clamp target, following administration of MK-1092 SC or glargine SC was determined by use of a continuous glucose infusion during the euglycemic clamp so that glucose levels remained in the euglycemic range and hypoglycemia was prevented. Blood glucose was monitored frequently (~every 5 minutes), allowing rapid changes to the rate of glucose infusion in Part 4 only. TWA(GIR)= Time-weighted average based on GIR values calculated as AUC (area under the curve) based on GIR values observed from time zero to t divided by t, t= 24 hours. Mean and 95% CI were based on a linear mixed effects model containing a fixed effect for treatment (MK, Glargine), period (Period 1, Period 2 and Period 3), a nested effect from participants within treatment, and interaction between treatment and period. MK-1092 or glargine was administered to a single cohort of participants in Periods 1, 2, and 3.
Time Frame: Up to approximately 24 hours post-dose
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: mg/kg/min
Groups:
- Part 4 (T2DM) MK-1092 32 Nmol/kg (Period 1): MK-1092, 8.0 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with T2DM
- Part 4 (T2DM) MK-1092 64 Nmol/kg (Period 3): MK-1092, 64 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with T2DM
- Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 1): Glargine 3.0 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with T2DM
- Part 1 (T2DM) Glargine 3.0 Nmol/kg (Period 2); Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 3): Glargine, 3.0 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with T2DM
Arm/Group | Part 4 (T2DM) MK-1092 32 Nmol/kg (Period 1) | Part 4 (T2DM) MK-1092 16 Nmol/kg (Period 2) | Part 4 (T2DM) MK-1092 64 Nmol/kg (Period 3) | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 1) | Part 1 (T2DM) Glargine 3.0 Nmol/kg (Period 2) | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 3)
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 3 | 3
mg/kg/min | 1.02 [0.83 to 1.21] | 0.78 [0.59 to 0.97] | 1.70 [1.51 to 1.89] | 0.50 [0.23 to 0.77] | 0.64 [0.37 to 0.91] | 0.67 [0.40 to 0.94]

9. Secondary Outcome: Maximal Plasma MK-1092 Concentration (Cmax) Parts 1 and 3
Description: Cmax is a measure of the maximum amount of drug in the plasma after the dose is given in Parts 1 and 3 only. The method of dispersion referenced below of geometric coefficient of variation is actually percent geometric coefficient of variation.
Time Frame: -15 min (predose), 10 min, 30 min, 1.0 hr, 1.5 hr, 2.0 hr, 3.0 hr, 4.0 hr, 6.0 hr, 9.0 hr, 12 hr, 18 hr, 24 hr, an additional sample will be collected at the end of the clamp, 2d, 3d, 4d, 5d and 7d after SC dose and at post-trial (Day 14 and Day 28)
Population: The analysis population included participants in Parts 1 and 3 who received MK-1092 and complied with the protocol sufficiently to ensure that data were likely to exhibit the effects of treatment, per the underlying scientific model. Compliance included exposure to treatment, availability of measurements, and absence of major protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Groups:
- Part 3 (T1DM) MK-1092 8.0 Nmol/kg: MK-1092 8.0 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with T1DM
Arm/Group | Part 1 (Healthy Adults) MK-1092 4.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 8.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 16 Nmol/kg | Part 1 (Healthy Adults) MK-1092 32 Nmol/kg | Part 1 (Healthy Adults) MK-1092 64 Nmol/kg | Part 3 (T1DM) MK-1092 8.0 Nmol/kg | Part 3 (T1DM) MK-1092 32 Nmol/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
nM | 0.382 (21.7) | 0.747 (25.0) | 1.63 (12.7) | 2.91 (18.7) | 6.82 (27.6) | 0.788 (20.4) | 3.43 (18.4)

10. Secondary Outcome: Area Under the Plasma Drug Curve From 0 to Infinity (AUC0-inf) MK-1092 Parts 1 and 3
Description: AUC0-inf is a measure of the total concentration levels of drug in the plasma after the dose is given in Parts 1 and 3 only. The method of dispersion referenced below of geometric coefficient of variation is actually percent geometric coefficient of variation.
Time Frame: as for outcome 9
Population: The analysis population included participants in Parts 1 & 3 who received MK-1092 and complied with the protocol (exposure to treatment, availability of measurements, absence of major protocol deviations) so that data exhibited effects of treatment. For the MK-1092 4.0 nmol/kg group, 5 participants were excluded (insufficient terminal phase data).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*hr
Arm/Group | Part 1 (Healthy Adults) MK-1092 4.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 8.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 16 Nmol/kg | Part 1 (Healthy Adults) MK-1092 32 Nmol/kg | Part 1 (Healthy Adults) MK-1092 64 Nmol/kg | Part 3 (T1DM) MK-1092 8.0 Nmol/kg | Part 3 (T1DM) MK-1092 32 Nmol/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6 | 6 | 6
nM*hr | 10.6 (NA) — Datum from only one participant was available so there is no associated percent geometric coefficient of variation. | 17.2 (12.0) | 37.5 (11.5) | 76.0 (10.2) | 161 (14.1) | 21.5 (22.2) | 74.9 (30.5)

11. Secondary Outcome: Rate of Plasma Drug Removal (CL/F) MK-1092 Parts 1 and 3
Description: CL/F is the rate at which a drug is removed from the body via renal, hepatic, and other clearance pathways after the dose is given in Parts 1 and 3 only. The method of dispersion referenced below of geometric coefficient of variation is actually percent geometric coefficient of variation.
Time Frame: as for outcome 9
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Groups:
- Part 3 (T1DM) MK-1092 8.0 Nmol/kg: Part 3 (Type 1 Diabetes Mellitus) MK-1092 8.0 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with T1DM
Arm/Group | Part 1 (Healthy Adults) MK-1092 4.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 8.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 16 Nmol/kg | Part 1 (Healthy Adults) MK-1092 32 Nmol/kg | Part 1 (Healthy Adults) MK-1092 64 Nmol/kg | Part 3 (T1DM) MK-1092 8.0 Nmol/kg | Part 3 (T1DM) MK-1092 32 Nmol/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6 | 6 | 6
L/hr | 25.6 (NA) — Datum from only one participant was available so there is no associated percent geometric coefficient of variation. | 35.0 (13.3) | 33.8 (19.8) | 32.2 (16.1) | 31.7 (13.9) | 33.6 (28.1) | 35.9 (26.6)

12. Secondary Outcome: Time to Reach Maximum Plasma MK-1092 Concentration (Tmax) Parts 1 and 3
Description: Tmax is the amount of the time to reach the maximum concentration in the plasma after the drug dose is given in Parts 1 and 3 only.
Time Frame: -15 min (predose), 10 min, 30 min, 1.0 hr, 1.5 hr, 2.0 hr, 3.0 hr, 4.0 hr, 6.0 hr, 9.0 hr, 12 hr, 18 hr, 24 hr, an additional sample will be collected and at the end of the clamp, 2d, 3d, 4d, 5d and 7d after SC dose and at post-trial (Day 14 and Day 28)
Population: as for outcome 9
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1 (Healthy Adults) MK-1092 4.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 8.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 16 Nmol/kg | Part 1 (Healthy Adults) MK-1092 32 Nmol/kg | Part 1 (Healthy Adults) MK-1092 64 Nmol/kg | Part 3 (T1DM) MK-1092 8.0 Nmol/kg | Part 3 (T1DM) MK-1092 32 Nmol/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hours | 18.00 [9.00 to 18.00] | 12.00 [4.00 to 18.00] | 18.00 [4.0 to 24.00] | 18.00 [9.00 to 18.00] | 12.00 [12.00 to 18.00] | 15.00 [9.00 to 18.00] | 15.04 [9.00 to 18.00]

13. Secondary Outcome: Time to Reach a 50% Decrease In Plasma MK-1092 Concentration (t1/2) Parts 1 and 3
Description: t1/2 is the time required for a given drug concentration in the plasma to decrease by 50% after the drug dose is given in Parts 1 and 3 only. The method of dispersion referenced below of geometric coefficient of variation is actually percent geometric coefficient of variation.
Time Frame: as for outcome 12
Population: The analysis population included participants in Parts 1 and 3 who received MK-1092 and complied with the protocol (treatments, measurements, major protocol deviations) so that data exhibited effects of treatment. For the MK-1092 4.0 and 64 nmol/kg groups, 5 and 1 participants, respectively, were excluded (insufficient terminal phase data).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1 (Healthy Adults) MK-1092 4.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 8.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 16 Nmol/kg | Part 1 (Healthy Adults) MK-1092 32 Nmol/kg | Part 1 (Healthy Adults) MK-1092 64 Nmol/kg | Part 3 (T1DM) MK-1092 8.0 Nmol/kg | Part 3 (T1DM) MK-1092 32 Nmol/kg
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 5 | 6 | 6
Hours | 6.39 (NA) — Datum from only one participant was available so there is no associated percent geometric coefficient of variation. . | 6.17 (29.3) | 5.41 (28.7) | 5.84 (16.5) | 9.27 (71.1) | 8.54 (23.2) | 6.70 (31.4)

14. Secondary Outcome: Maximal Plasma MK-1092 Concentration (Cmax) Part 4
Description: Cmax is a measure of the maximum amount of drug in the plasma after the dose is given in Parts 4 only. The method of dispersion referenced below of geometric coefficient of variation is actually percent geometric coefficient of variation.
Time Frame: as for outcome 9
Population: The analysis population included participants in Part 4 who received MK-1092 and complied with the protocol sufficiently to ensure that data were likely to exhibit the effects of treatment, per the underlying scientific model. Compliance included exposure to treatment, availability of measurements, and absence of major protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Part 4 (T2DM) MK-1092 32 Nmol/kg (Period 1) | Part 4 (T2DM) MK-1092 16 Nmol/kg (Period 2) | Part 4 (T2DM) MK-1092 64 Nmol/kg (Period 3)
Number analyzed (Participants) | 6 | 6 | 6
nM | 1.72 (46.0) | 1.14 (32.6) | 3.60 (23.0)

15. Secondary Outcome: Area Under the Plasma Drug Curve From 0 to Infinity (AUC0-inf) MK-1092 Part 4
Description: AUC0-inf is a measure of the total concentration levels of drug in the plasma after the dose is given in Part 4 only. The method of dispersion referenced below of geometric coefficient of variation is actually percent geometric coefficient of variation.
Time Frame: as for outcome 9
Population: The analysis population included participants in Part 4 who received MK-1092 and complied with the protocol (exposure to treatment, measurement availability, major protocol deviations) so that data exhibited effects of treatment. Seven participants (Period 1:1; Period 2:3; Period 3:3) were excluded due to insufficient terminal phase data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*hr
Arm/Group | Part 4 (T2DM) MK-1092 32 Nmol/kg (Period 1) | Part 4 (T2DM) MK-1092 16 Nmol/kg (Period 2) | Part 4 (T2DM) MK-1092 64 Nmol/kg (Period 3)
Number analyzed (Participants) | 5 | 3 | 3
nM*hr | 46.1 (34.4) | 32.7 (48.8) | 111 (20.7)

16. Secondary Outcome: Rate of Plasma Drug Removal (CL/F) MK-1092 Part 4
Description: CL/F is the rate at which a drug is removed from the body via renal, hepatic, and other clearance pathways after the dose is given in Part 4 only. The method of dispersion referenced below of geometric coefficient of variation is actually percent geometric coefficient of variation.
Time Frame: as for outcome 9
Population: The analysis population included participants in Parts 4 who received MK-1092 and complied with the protocol (exposure to treatment, measurement availability, major protocol deviations) so that data exhibited effects of treatment. Seven participants (Period 1:1; Period 2:3; Period 3:3) were excluded due to insufficient terminal phase data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Part 4 (T2DM) MK-1092 32 Nmol/kg (Period 1) | Part 4 (T2DM) MK-1092 16 Nmol/kg (Period 2) | Part 4 (T2DM) MK-1092 64 Nmol/kg (Period 3)
Number analyzed (Participants) | 5 | 3 | 3
L/hr | 55.6 (27.4) | 45.9 (52.5) | 40.7 (13.5)

17. Secondary Outcome: Time to Reach Maximum Plasma MK-1092 Concentration (Tmax) Part 4
Description: Tmax is the amount of the time to reach the maximum concentration in the plasma after the drug dose is given in Part 4 only.
Time Frame: as for outcome 12
Population: as for outcome 14
Measure: Median (Full Range); unit: Hours
Groups:
- Part 4 (T2MD) MK-1092 64 Nmol/kg (Period 3): MK-1092, 64 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with T2DM
Arm/Group | Part 4 (T2DM) MK-1092 32 Nmol/kg (Period 1) | Part 4 (T2DM) MK-1092 16 Nmol/kg (Period 2) | Part 4 (T2MD) MK-1092 64 Nmol/kg (Period 3)
Number analyzed (Participants) | 6 | 6 | 6
Hours | 14.99 [9.00 to 18.00] | 18.00 [12.00 to 18.00] | 21.04 [18.00 to 24.00]

18. Secondary Outcome: Time to Reach a 50% Decrease In Plasma MK-1092 Concentration (t1/2) Part 4
Description: t1/2 is the time required for a given drug concentration in the plasma to decrease by 50% after the drug dose is given in Part 4 only. The method of dispersion referenced below of geometric coefficient of variation is actually percent geometric coefficient of variation.
Time Frame: as for outcome 12
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 4 (T2DM) MK-1092 32 Nmol/kg (Period 1) | Part 4 (T2DM) MK-1092 16 Nmol/kg (Period 2) | Part 4 (T2DM) MK-1092 64 Nmol/kg (Period 3)
Number analyzed (Participants) | 5 | 3 | 3
Hours | 8.26 (39.1) | 9.09 (20.4) | 7.28 (30.6)

19. Secondary Outcome: Maximal Plasma Insulin Glargine Concentration (Cmax) Parts 1 and 3
Description: Cmax is a measure of the maximum amount of drug in the plasma after the dose is given in Parts 1 and 3 only. Healthy participants received glargine in Panel A-E, and participants with T1DM received glargine in Panel G and H. The method of dispersion referenced below of geometric coefficient of variation is actually percent geometric coefficient of variation. In Part 1, 9 participants (across 5 dosing panels) received glargine and had quantifiable glargine levels, and, in Part 3, 4 participants (across 2 dosing panels) received glargine and had quantifiable glargine levels. These 9 participants in Part 1 were analyzed together and these 4 participants in Part 3 were analyzed together given the small numbers and same treatment (same dose of glargine) received.
Time Frame: as for outcome 9
Population: The analysis population included participants in Parts 1 and 3 who received glargine and complied with the protocol sufficiently so that the data exhibited effects of treatment. One participant (Part 1) was excluded (no quantifiable glargine concentration). Data across panels were pooled for Parts 1 and 3.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Part 1 (Healthy Adults) Glargine 3.0 Nmol/kg | Part 3 (T1DM) Glargine 3.0 Nmol/kg
Number analyzed (Participants) | 9 | 4
pg/mL | 115 (48.4) | 186 (33.8)

20. Secondary Outcome: Area Under the Plasma Drug Curve From 0 to Infinity (AUC0-inf) Insulin Glargine Parts 1 and 3
Description: AUC0-inf is a measure of the total concentration levels of drug in the plasma after the dose is given in Parts 1 and 3 only. Healthy participants received glargine in Panel A-E, and participants with T1DM received glargine in Panel G and H. The method of dispersion referenced below of geometric coefficient of variation is actually percent geometric coefficient of variation. In Part 1, 8 participants (across 5 dosing panels) received glargine and had sufficient terminal phase data, and, in Part 3, 3 participants (across 2 dosing panels) received glargine and had sufficient terminal phase data. These 8 participants in Part 1 were analyzed together and these 3 participants in Part 3 were analyzed together given the small numbers and same treatment (same dose of glargine) received.
Time Frame: as for outcome 9
Population: The analysis population included participants in Parts 1 and 3 who received glargine and complied with the protocol sufficiently so that the data exhibited the effects of treatment. Two participants in Part 1 and 1 in Part 3 were excluded due to insufficient terminal phase data. Data across panels were pooled for Parts 1 and 3.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*pg/mL
Groups:
- Part 3 (T1DM) Glargine 3.0 Nmol/kg: Glargine 3.0 nmol/kg, SC, as a single dose under the euglycemic clamp in participants with T1DM
Arm/Group | Part 1 (Healthy Adults) Glargine 3.0 Nmol/kg | Part 3 (T1DM) Glargine 3.0 Nmol/kg
Number analyzed (Participants) | 8 | 3
hr*pg/mL | 3180 (44.7) | 4240 (93.9)

21. Secondary Outcome: Time to Reach Maximum Plasma Insulin Glargine Concentration (Tmax) Parts 1 and 3
Description: Tmax is the amount of the time to reach the maximum concentration in the plasma after the drug dose is given in Parts 1 and 3 only. Healthy participants received glargine in Panel A-E, and participants with T1DM received glargine in Panel G and H. In Part 1, 9 participants (across 5 dosing panels) received glargine and had quantifiable glargine levels, and, in Part 3, 4 participants (across 2 dosing panels) received glargine and had quantifiable glargine levels. These 9 participants in Part 1 were analyzed together and these 4 participants in Part 3 were analyzed together given the small numbers and same treatment (same dose of glargine) received.
Time Frame: as for outcome 12
Population: The analysis population included participants in Parts 1 and 3 who received glargine and complied with the protocol so that data likely exhibited effects of treatment. One participant (Part 1) was excluded (no quantifiable glargine concentration). Data across panels were pooled for Parts 1 and 3.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1 (Healthy Adults) Glargine 3.0 Nmol/kg | Part 3 (T1DM) Glargine 3.0 Nmol/kg
Number analyzed (Participants) | 9 | 4
Hours | 1.98 [0.48 to 11.97] | 1.74 [0.5 to 3.00]

22. Secondary Outcome: Time to Reach a 50% Decrease In Plasma Insulin Glargine Concentration (t1/2) Parts 1 and 3
Description: t1/2 is the time required for a given drug concentration in the plasma to decrease by 50% after the drug dose is given in Parts 1 and 3 only. Healthy participants received glargine in Panel A-E, and participants with T1DM received glargine in Panel G and H. The method of dispersion referenced below of geometric coefficient of variation is actually percent geometric coefficient of variation. In Part 1, 8 participants (across 5 dosing panels) received glargine and had sufficient terminal phase data, and, in Part 3, 3 participants (across 2 dosing panels) received glargine and sufficient terminal phase data. These 8 participants in Part 1 were analyzed together and these 3 participants in Part 3 were analyzed together given the small numbers and same treatment (same dose of glargine) received.
Time Frame: as for outcome 12
Population: The analysis population included participants in Parts 1 and 3 who received glargine and sufficiently complied with the protocol so that the data exhibited the effects of treatment. Two participants excluded in Part 1 and 1 participant excluded in Part 3 due to insufficient terminal phase data. Data across panels were pooled for Parts 1 and 3.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1 (Healthy Adults) Glargine 3.0 Nmol/kg | Part 3 (T1DM) Glargine 3.0 Nmol/kg
Number analyzed (Participants) | 8 | 3
Hours | 18.8 (64.5) | 15.0 (65.8)

23. Secondary Outcome: Maximal Plasma Insulin Glargine Concentration (Cmax) Part 4
Description: as for outcome 14
Time Frame: as for outcome 9
Population: The analysis population included participants in Part 4 who received glargine and complied with the protocol sufficiently to ensure that data were likely to exhibit the effects of treatment, per the underlying scientific model. Compliance included exposure to treatment, availability of measurements, and absence of major protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 1) | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 2) | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 3)
Number analyzed (Participants) | 3 | 3 | 3
pg/mL | 85.6 (18.0) | 91.9 (35.1) | 105 (33.9)

24. Secondary Outcome: Area Under the Plasma Drug Curve From 0 to Infinity (AUC0-inf) Insulin Glargine Part 4
Description: as for outcome 15
Time Frame: as for outcome 9
Population: The analysis population included participants in Part 4 who received glargine and complied with the protocol (exposure to treatment, availability of measurements, major protocol deviations) so that data exhibited effects of treatment. Five participants (Period 1:1; Period 2:2; Period 3:2) were excluded due to insufficient terminal phase data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*pg/mL
Arm/Group | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 1) | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 2) | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 3)
Number analyzed (Participants) | 2 | 1 | 1
hr*pg/mL | 4960 (66.2) | 928 (NA) — Datum from only one participant was available so there is no associated geometric coefficient of variation. | 8020 (NA) — Datum from only one participant was available so there is no associated geometric coefficient of variation.

25. Secondary Outcome: Time to Reach Maximum Plasma Insulin Glargine Concentration (Tmax) Part 4
Description: as for outcome 17
Time Frame: -15 min (predose), 10 min, 30 min, 1.0 hr, 1.5 hr, 2.0 hr, 3.0 hr, 4.0 hr, 6.0 hr, 9.0 hr, 12 hr, 18 hr, 24 hr, an additional sample will be collected and at the end of the clamp, 2d, 3d, 4d, 5d and 7d after SC dose and at post-trial (Day 14 and Day 28) ]
Population: as for outcome 23
Measure: Median (Full Range); unit: Hr
Arm/Group | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 1) | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 2) | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 3)
Number analyzed (Participants) | 3 | 3 | 3
Hr | 1.00 [0.98 to 11.98] | 2.00 [1.00 to 9.00] | 2.98 [1.00 to 11.98]

26. Secondary Outcome: Time to Reach a 50% Decrease In Plasma Insulin Glargine Concentration (t1/2) Part 4
Description: as for outcome 18
Time Frame: as for outcome 25
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 1) | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 2) | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 3)
Number analyzed (Participants) | 2 | 1 | 1
Hours | 45.2 (53.2) | 8.10 (NA) — Datum from only one participant was available so there is no associated geometric coefficient of variation. | 46.5 (NA) — Data from only one participant was available so there is no associated geometric coefficient of variation.

ADVERSE EVENTS:
Time Frame: Up to 112 days
Description: Post-trial adverse events were pooled across the arms in each part of the study. Adverse events that occurred beyond 14 days of dosing were considered Post-Trial AEs. Given the half-life of MK-1092 and glargine, any events observed beyond 14 days would not be considered a result of study drug and were therefore presented together.
Groups:
- Part 1 (Healthy Adults) Post-trial: Glargine or MK-1091 as a single dose under the euglycemic clamp in healthy adults in the Post-trial period
- Part 2 (Healthy Adults) MK-1092 + Insulin Lipro Post-trial: MK-1092, 8.0 nmol/kg selection based on Part 2 + Insulin lipro (Humalog®), 1.2 nmol/kg, as a single dose under the euglycemic clamp in healthy participants in the Post-trial period
- Part 3 (T1DM) Glargine 3.0 Nmol/kg: Glargine 3.0 nmol/kg SC as a single dose under euglycemic clamp in participants with T1DM
- Part 3 (T1DM) MK-1092 8.0 Nmol/kg: MK-1092 8.0 nmol/kg SC as a single dose under euglycemic clamp in participants with T1DM
- Part 3 (T1DM) MK-1092 32 Nmol/kg: MK-1092 32 nmol/kg SC as a single dose under euglycemic clamp in participants with T1DM
- Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 1): Glargine 3.0 nmol/kg, SC, as a single dose under euglycemic clamp in participants with T1DM in Period 1
- Part 4 (T2DM) 64 Nmol/kg (Period 3): MK-1092, 64 nmol/kg dose as a single dose under euglycemic clamp in participants with T2DM
- Part 4 (T2DM) Post-Trial: Glargine or MK-1092 as a single dose under euglycemic clamp in participants with T2DM in the Post-trial period
Arm/Group | Part 1 (Healthy Adults) Glargine 3.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 4.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 8.0 Nmol/kg | Part 1 (Healthy Adults) MK-1092 16 Nmol/kg | Part 1 (Healthy Adults) MK-1092 32 Nmol/kg | Part 1 (Healthy Adults) MK-1092 64 Nmol/kg | Part 1 (Healthy Adults) Post-trial | Part 2 (Healthy Adults) MK-1092 + Insulin Lipro | Part 2 (Healthy Adults) MK-1092 + Insulin Lipro Post-trial | Part 3 (T1DM) Glargine 3.0 Nmol/kg | Part 3 (T1DM) MK-1092 8.0 Nmol/kg | Part 3 (T1DM) MK-1092 32 Nmol/kg | Part 3 (T1DM) Post-trial | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 1) | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 2) | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 3) | Part 4 (T2DM) MK-1092 32 Nmol/kg (Period 1) | Part 4 (T2DM) MK-1092 16 Nmol/kg (Period 2) | Part 4 (T2DM) 64 Nmol/kg (Period 3) | Part 4 (T2DM) Post-Trial
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/40 | 0/4 | 0/4 | 0/4 | 0/6 | 0/6 | 0/16 | 0/3 | 0/3 | 0/3 | 0/6 | 0/6 | 0/6 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/40 | 0/4 | 0/4 | 0/4 | 0/6 | 0/6 | 0/16 | 0/3 | 0/3 | 0/3 | 0/6 | 0/6 | 0/6 | 0/9
Other Adverse Events (participants affected / at risk) | 1/10 | 1/6 | 4/6 | 3/6 | 3/6 | 2/6 | 0/40 | 3/4 | 1/4 | 2/4 | 6/6 | 5/6 | 2/16 | 3/3 | 1/3 | 0/3 | 3/6 | 3/6 | 4/6 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 (Healthy Adults) Glargine 3.0 Nmol/kg (N=10) | Part 1 (Healthy Adults) MK-1092 4.0 Nmol/kg (N=6) | Part 1 (Healthy Adults) MK-1092 8.0 Nmol/kg (N=6) | Part 1 (Healthy Adults) MK-1092 16 Nmol/kg (N=6) | Part 1 (Healthy Adults) MK-1092 32 Nmol/kg (N=6) | Part 1 (Healthy Adults) MK-1092 64 Nmol/kg (N=6) | Part 1 (Healthy Adults) Post-trial (N=40) | Part 2 (Healthy Adults) MK-1092 + Insulin Lipro (N=4) | Part 2 (Healthy Adults) MK-1092 + Insulin Lipro Post-trial (N=4) | Part 3 (T1DM) Glargine 3.0 Nmol/kg (N=4) | Part 3 (T1DM) MK-1092 8.0 Nmol/kg (N=6) | Part 3 (T1DM) MK-1092 32 Nmol/kg (N=6) | Part 3 (T1DM) Post-trial (N=16) | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 1) (N=3) | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 2) (N=3) | Part 4 (T2DM) Glargine 3.0 Nmol/kg (Period 3) (N=3) | Part 4 (T2DM) MK-1092 32 Nmol/kg (Period 1) (N=6) | Part 4 (T2DM) MK-1092 16 Nmol/kg (Period 2) (N=6) | Part 4 (T2DM) 64 Nmol/kg (Period 3) (N=6) | Part 4 (T2DM) Post-Trial (N=9)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Administration site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site dermatitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 6 (11) | 3 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pseudohypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT03170544/Prot_SAP_000.pdf